CLINICAL TRIAL: NCT00533338
Title: Weight Gain Prevention for Breast Cancer Survivors
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Lance Armstrong Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2005-0888
Record Dates: First submitted 2007-09-19; First posted 2007-09-21 (Estimated); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Cancer Survivors; Weight Gain Prevention; Diet; Exercise; Questionnaire; Survey
MeSH Terms: conditions — Breast Neoplasms; Motor Activity | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Weight Gain Prevention Program (Experimental): Intervention program including in-person instruction and counseling about exercise and diet, exercise practice sessions, and telephone counseling. Packet of questionnaires will be completed.
  Interventions: Behavioral: Weight Gain Prevention Program; Behavioral: Questionnaire
- Standard Care Group (Active Comparator): Packet of questionnaires will be completed.
  Interventions: Behavioral: Questionnaire

INTERVENTIONS:
Behavioral: Weight Gain Prevention Program — Intervention program including in-person instruction and counseling about exercise and diet, exercise practice sessions, and telephone counseling.
  Arms: Weight Gain Prevention Program
Behavioral: Questionnaire — Packet of questionnaires will be completed.
  Other Names: Survey

SUMMARY:
The specific aims of this study are:

1. To test the feasibility of a randomized controlled trial of a weight gain prevention program for breast cancer survivors that combines exercise and dietary changes during treatment. Feasibility will be evaluated by examining data on recruitment rate, attendance at intervention sessions, drop-out rates in both study conditions, assessment completion rates, and participant feedback.
2. To test the effect of a weight gain prevention program, compared to usual care, on weight, body composition, and biomarkers related to breast cancer prognosis.
3. To explore whether changes in physical activity, energy intake, and resting energy expenditure predict weight gain among breast cancer survivors.
4. To test the effect of a weight gain prevention program on quality of life variables.

DETAILED DESCRIPTION:
Women who are breast cancer patients having chemotherapy before surgery will be invited to participate in the study. You will be allowed to participate in this study only if your physician feels it is safe for you to participate in moderate physical activity, so you will be asked to have him or her complete a form about your health conditions. Information about the cancer and your treatment history will be obtained from your medical records as part of the study.

If you agree to take part in this study, you will asked to come in for 2 visits at the beginning of the study. At your first visit, your resting energy expenditure (REE) will be measured. To test your REE, you will lie down on a bed while wearing a mask to measure the air you let out when you breathe. You will have an electrocardiogram (ECG -- a test that measures the electrical activity of the heart). Blood (about 2 teaspoons) will be drawn to measure biomarkers, that may affect breast cancer. You will receive a packet of quality of life questionnaires which will take 45 minutes to complete. You will also receive an actigraph (a small, light-weight device that is worn on the waist during the day) that provides researchers with information on your physical activity. You will be asked to wear the actigraph for 7 days before your second visit. You will be given a diet questionnaire to complete at home. The diet questionnaire will take 60 minutes to complete. You will be asked to bring the actigraph and questionnaires to a baseline study visit.

At the second study visit you will also complete questionnaires about your physical activity.

Your blood pressure and heart rate will be measured. Your physical fitness will be checked by an exercise test done on a treadmill. The exercise test will be monitored by a qualified health care provider and performed by a certified exercise specialist with training in emergency procedures. The exercise intensity will begin at a low level and will be increased over time. The test may be stopped at any time if you experience signs of fatigue or changes in your heart rate, ECG, or blood pressure. You may also stop the test whenever you wish.

Your height, weight, skinfolds, and hip and waist circumference will be measured. Your arm, shoulder, and leg strength will be checked by asking you to stand on a platform and grasp a bar connected to a strain gauge that measures force. Your hip and lower back flexibility will checked using a 'sit and reach' method. Flexibility in your arm will be checked using a goniometer, a small plastic measuring device similar to a ruler.

You will be given a packet of 10 collection tubes for collecting saliva samples with instruction on collecting the samples over 2 days during the next week. You will also be given a special mailer with which to return the samples. The second study visit will take about 2 hours.

After your initial visit, you will be asked to come to M. D. Anderson to complete a Dual energy x-ray absorptiometry (DEXA) scan to evaluate body composition.

At your baseline study visit, you will be randomly assigned (as in the toss of a coin) to either a weight gain prevention group or a standard of care group. An equal number of people will be assigned to each group.

If you are assigned to the intervention group, you will attend individual in-person study visits at M. D. Anderson to receive instruction and counseling about exercise and diet.

While you are receiving chemotherapy, you will attend 1, 60-minute study visit per week for 16 weeks. During these visits, you will be given instructions on resistance and flexibility exercises, using a pedometer (a small device that is worn during the day to give you information about the number of steps you take), and making changes in your diet. You will practice the exercises during this session, and receive feedback. Some of these session might be video taped. You will be asked to give permission for the videotaping before the session begins.

After the 16 weeks of in-person sessions, you will receive 1 telephone counseling session per week for the remainder of the time you are on chemotherapy. Each telephone call will take about 15-20 minutes. Some of these sessions might be tape-recorded. You will be asked permission to tape-record the session before the telephone counseling session is begun. You will receive written materials about making changes to your diet and exercise behavior. The written materials will have information about overcoming barriers, rewarding yourself, and time management. You will also receive hand weights, a step, and a stability ball for exercising at home and a pedometer for monitoring your walking. The hand weights, step, stability ball, and pedometer will be yours to keep. Based on the strength assessment, tailored resistance exercises will be prescribed. You will do the exercises up to 3 times per week. The exercise will target the major muscle groups.

After you have recovered from surgery, you will have 1 study visit a week for 3 weeks. You will practice the exercises and again receive counseling to encourage you to exercise and to eat according to your dietary recommendations. The exercises may be modified at this visit, if necessary.

After these 3 weeks, you will receive 1 phone call a week for the next 6 weeks. Each telephone call will take about 15-20 minutes. You will also receive additional written materials that will include exercises and recommendations for maintaining the behavioral changes made.

Regardless of which group you are in, you will be asked to come to M. D. Anderson for follow-up assessments at the mid-point and end of chemotherapy, after recovering from surgery, then 9 weeks and 6 months after surgery. You will be asked to come to M. D. Anderson to complete a DEXA scan to evaluate body composition and bone mineral density at the end of chemotherapy. For safety purposes, researchers will look for lymphedema at follow-up evaluations after recovering from surgery, then 9 weeks and 6 months after surgery. About 8 days before each follow-up visit we will send you a packet of seven questionnaires that will take 45 minutes to complete, and an actigraph. You will be called on the day you are supposed to wear the actigraph, and you will be given instructions about completing the questionnaires. You will bring the questionnaires and actigraph to your study visits. You will have the same tests and procedures at these study visits as you had at the baseline visit.

You will be considered off-study 6 months after your surgery.

This is an investigational study. About 60 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Woman with newly diagnosed stage II or III breast cancer.
2. Over 18 years of age.
3. Beginning neo-adjuvant chemotherapy at M. D. Anderson (no more than 3 weeks from the administration of the first cycle).
4. Speaks and reads English.
5. Oriented to person, place, and time.
6. Able to come to M. D. Anderson once a week for intervention.
7. Has physician clearance to engage in moderate physical activity.
8. Lives in Harris County, Texas or a county contiguous to Harris County, Texas.

Exclusion Criteria:

1. Have any of the following conditions defined by the American College of Sports Medicine as absolute contraindications to exercise testing (a recent significant change in the resting ECG suggesting significant ischemia, recent myocardial infarction (within 2 days) or acute cardiac event; unstable angina; uncontrolled cardiac arrhythmias causing symptoms or hemodynamic compromise; severe symptomatic aortic stenosis; uncontrolled symptomatic heart failure; acute pulmonary embolus or pulmonary infarction; acute myocarditis or pericarditis; suspected or known dissecting aneurysm; acute infection).
2. Have any of the following conditions as defined by the American College of Sports Medicine as relative contraindications to exercise testing (left main coronary stenosis; moderate stenotic valvular heart disease; electrolyte abnormalities; severe arterial hypertension at rest; hypertrophic cardiomyopathy and other forms of outflow tract obstruction; neuromuscular, musculoskeletal, or rheumatoid disorders that are exacerbated by exercise; high-degree atrioventricular block; ventricular aneurysm; uncontrolled metabolic disease; chronic infectious disease).
3. Right or left bundle branch block.
4. Baseline ST segment or T wave changes that would make monitoring of the ECG stress test indeterminate.
5. Uncontrolled asthma.
6. Have other medical contraindications as defined by the patient's physician.
7. Have inflammatory breast cancer.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2007-07-20 (Actual); Primary Completion 2020-07-31 (Estimated); Study Completion 2020-07-31 (Estimated)

PRIMARY OUTCOMES:
Weight or Percentage (%) Body Fat | Six assessments: baseline, 3 months after starting chemotherapy, at the end of chemotherapy, after recovery from surgery, at the end of the 9-week booster intervention, and 6 months after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Karen Basen-Engquist, PhD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Basen-Engquist KM, Raber M, Carmack CL, Arun B, Brewster AM, Fingeret M, Schembre SM, Harrison C, Perkins HY, Li Y, Song J, Chen M, Murray JL. Feasibility and efficacy of a weight gain prevention intervention for breast cancer patients receiving neoadjuvant chemotherapy: a randomized controlled pilot study. Support Care Cancer. 2020 Dec;28(12):5821-5832. doi: 10.1007/s00520-020-05411-2. Epub 2020 Apr 5. PMID 32249355
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org